CLINICAL TRIAL: NCT00356044
Title: Femoral Versus Radial Access for Coronary Intervention in the Acute Phase of ST-Elevation Myocardial Infarction
Brief Title: Arterial Access for Coronary Intervention in Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Juan Canalejo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEICG 2004/063
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2007-07-11 (Estimated); Status verified 2007-07

CONDITIONS: Myocardial Infarction; Angioplasty, Transluminal, Percutaneous Coronary; Myocardial Reperfusion
Keywords: Transradial access; Femoral access; Femoral vs radial access
MeSH Terms: conditions — Myocardial Infarction | interventions — Angioplasty, Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Coronary angioplasty

SUMMARY:
The aim of this study is to compare the radial and femoral access for percutaneous interventions in the acute phase of the ST elevation acute myocardial infarction in terms of efficacy and security.

DETAILED DESCRIPTION:
Some groups have previously used the radial artery as the access route in the procedures of percutaneous coronary revascularization, with good results. The advantages of the radial compared with femoral access are related to a lower incidence of vascular complications. The radial access has also inconveniences such as a less predictable anatomy which can make the procedure difficult and prolong the time required.The patients with ST elevation myocardial infarction have an increased risk of vascular complications after interventional procedures because previous antithrombotic or thrombolytic therapy.On the other hand, the time and success of the procedure are significant prognostic issues.In this sitting, the radial approach might reduce vascular complications and increase other cardiovascular events when comparing with the classical femoral access. For this reason, the purpose of the study is to compare both arterial access in terms of efficacy and security and to quantify the consequences of the advantages and drawbacks of both.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ST elevation acute myocardial infarction referred for primary,facilitated or of rescue coronary angioplasty in the first 12 hours since the start of the symptoms.

Exclusion Criteria:

* Patients in cardiogenic shock were excluded following operator criteria.
* Previous coronary surgery with mammary artery graft
* Coronary artery intervention in the previous month
* Absolute or relative contraindication for access via the radial artery route:Radial pulse absent or weak, abnormal Allen test,anatomy known to impede the use of the radial route or hemodialysis or advanced chronic renal insufficiency (creatinine >3 mg/dl).
* Patients with absolute or relative contraindication for the use of the femoral route.
* Absence of informed consent from the patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2004-05; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
All cause mortality at 30 days | within the first 30 days (plus or minus 5 days) after the index myocardial infarction
New ST elevation acute myocardial infarction at 30 days | within the first 30 days (plus or minus 5 days) after the index myocardial infarction
Coronary revascularization as a result of recurrent ischemia at 30 days | within the first 30 days (plus or minus 5 days) after the index myocardial infarction
Major vascular complications at 30 days. | within the first 30 days (plus or minus 5 days) after the index myocardial infarction

SECONDARY OUTCOMES:
Embolic stroke at 30 days | within the first 30 days (plus or minus 5 days) after the index myocardial infarction
Coronary revascularization at 30 days | within the first 30 days (plus or minus 5 days) after the index myocardial infarction
Cardiovascular mortality at 30 days | within the first 30 days (plus or minus 5 days) after the index myocardial infarction
Procedural time
Hospital stay
Estimation of costs

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Vazquez-Rodriguez, MD, Study Chair — Hospital Juan Canalejo; Jose A Baz, Alonso, Principal Investigator — Hospital do meixoeiro; Andrés Iñiguez-Romo, MD, Study Director — Hospital do Meixoeiro; Nicolás Vázquez-González, MD, Study Director — Hospital Juan Canalejo; Ramón Calviño-Santos, MD, Principal Investigator — Hospital Juan Canalejo; Antonio Amaro-Cendón, MD, Study Director — Complejo Hospitalario Universitario de Santiago; Ramiro Trillo, Nouche, Principal Investigator — Complejo Hospitalario Universitario de Santiago
Locations (3):
- Spain (3):
  - Hospital Juan Canalejo, A Coruña, A Coruña
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital do Meixoeiro, Vigo, Pontevedra

REFERENCES:
- [Background] Saito S, Tanaka S, Hiroe Y, Miyashita Y, Takahashi S, Tanaka K, Satake S. Comparative study on transradial approach vs. transfemoral approach in primary stent implantation for patients with acute myocardial infarction: results of the test for myocardial infarction by prospective unicenter randomization for access sites (TEMPURA) trial. Catheter Cardiovasc Interv. 2003 May;59(1):26-33. doi: 10.1002/ccd.10493. PMID 12720237
- [Background] Exaire JE, Dauerman HL, Topol EJ, Blankenship JC, Wolski K, Raymond RE, Cohen EA, Moliterno DJ; TARGET Investigators. Triple antiplatelet therapy does not increase femoral access bleeding with vascular closure devices. Am Heart J. 2004 Jan;147(1):31-4. doi: 10.1016/j.ahj.2003.07.019. PMID 14691415
- [Result] Vazquez Rodriguez JM, Calvino Santos R, Baz Alonso JA, Trillo Nouche R, Salgado Fernandez J, Sanmartin Fernandez M, et al. Radial vs. Femoral access in emergent coronary interventions for acute myocerdial infarction with ST segment elevation (abstract). Innovation in Intervention: i2 Summit 2007 Abstract Sessions. 10.1016/j.jacc.2007.01.048. J Am Coll Cardiol 2007;49(9_Suppl_B):12B.